CLINICAL TRIAL: NCT02340559
Title: Effectiveness of Meta-Cognitive Training (EMC) on Symptmos, Metacognition, Social and Neuropsychological Functioning in People With Psychosis of Brief Evolution
Brief Title: Effectiveness of Meta-Cognitive Training (EMC) in People With Psychosis of Brief Evolution.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: Parc Sanitari Sant Joan de Déu (Other); Corporacion Parc Tauli (Other); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); Fundación para la Investigación del Hospital Clínico de Valencia (Other); Centre d'Higiene Mental Les Corts (Other); Institut d´Assistència Sanitària Girona (Unknown); Servicio Andaluz de Salud de Granada, Málaga y Jaén (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI11/01347
Record Dates: First submitted 2015-01-13; First posted 2015-01-16 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Psychosis
Keywords: meta-cognition; positive symptoms; early phases; schizophrenia
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Meta-cognitive Training (Experimental): The metacognitive training program is comprised of eight modules targeting common cognitive errors in schizophrenia. The modules are : attributional distortions (module 1), a jumping to conclusions bias (module 2 and 7), a bias against disconfirmatory evidence (module 3), deficits in theory of mind (module 4 and 6), over-confidence in memory errors (module 5) and depressive cognitive patterns (module 8).
  The treatment group consist of 8 weekly sessions of 45-60 minutes with a total of 4 to 8 patients per group.
  Interventions: Behavioral: Psychoeducational group
- Psychoeducational group (Active Comparator): In the control group the modules worked were: 1. Healthy Habits, 2. Risk Behaviors, 3. Prevention of relapse, 4 and 5.Videoforum, 6. Resources of work and development of curriculum vitae 7. Leisure activities, and 8. Resources of the community. The psychoeducational group consist of 8 weekly sessions of 45-60 minutes with a total of 4 to 8 patients per group.
  Interventions: Behavioral: Meta-cognitive Training

INTERVENTIONS:
Behavioral: Meta-cognitive Training
  Arms: Psychoeducational group
Behavioral: Psychoeducational group
  Arms: Meta-cognitive Training

SUMMARY:
The purpose of this study is to assess the effectiveness of Meta-Cognitive Training (EMC) in people with a brief psychotic disorder, especially positive symptoms.

The secondary objectives would be to assess the effect of EMC on metacognition (cognitive distortions and deficits in theory of mind), psychosocial functioning and quality of life, neuropsychological functioning and gender, as well as determine the changes produced by EMC in the insight of each session and the maintenance of the effects of EMC program at six months of treatment.

DETAILED DESCRIPTION:
The study is a randomized clinical trial in which a group will receive the Meta-Cognitive Training (EMC) and a control group will receive a journal workshop.

The evaluator will be blind to the group that owns the patients included. The total simple will be of 122 people with a psychotic disorder, less than 5 years of evolution and a score at or above 3 on the PANSS during the last year. Patients should be attended in one of the next services: Parc Sanitari Sant Joan de Déu, Corporació Sanitària Parc Taulí, Hospital de la Santa Creu i Sant Pau, Hospital Clínic de Valencia, Centre d´Higiene Mental de les Corts, Institut d´Assitència Sanitària Girona, Servicio Andaluz de Granada, Málaga y Jaén. The assessment was performed at baseline, at the end of treatment and six month follow-up.

The assessment includes: psychopathology and insight ( PANSS, PSYRATS, PDI, GAF, BDI, BCIS, Sumd), meta-cognition (jumping to conclusions, IPSAQ, TCI), neuropsychology (WCST, TMT, CPT-II, TAVEC, WAIS) and social functioning and quality of life (EFS, DAS-SV, SLDS). The insight will be assessed at the final of each session (BCIS). The treatment and control group consist of 8 weekly sessions of 45-60 minutes with a total of 4 to 8 patients per group. The EMC group material is translated and validated in Spanish by investigators of the team.

The primary analysis variable is the difference between the scores of experimental and control group in the symptoms scales (especially positive). Secondary outcomes will change in other assessments of social functioning, metacognition (cognitive distortions and theory of mind) and neuropsychological variables. Were analyzed using regression and ANCOVA methods with SPSS 19.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of : schizophrenia, schizoaffective disorder, brief psychotic disorder, delusional disorder, schizophreniform disorder, psychotic disorder not otherwise specified.
* Less than 5 years of evolution.
* Score at or above 4 on the PANSS during the last year (delusions, grandiosity, suspiciousness).

Exclusion Criteria:

* Neurological disorder which impairs cognition.
* Intellectual Disability.
* Score at or above 5 on the PANSS ( Hostility and Uncooperativeness); score at or above 6 on the PANSS (suspiciousness).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2012-08; Primary Completion 2013-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
PANSS. Positive and Negative Syndrome Scale | baseline, 2 months (post-treatment) and 6 months of follow-up
  The Positive and Negative Syndrome Scale (PANSS)(Kay et al., 1987; Peralta and Cuesta, 1994) measures 30 symptoms on a scale of 1-7, with higher scores indicating greater psychopathology. The PANSS contains three sub-scales: positive, negative and general symptoms.
PSYRATS. Psychotic Symptoms Rating Scale | baseline, 2 months (post-treatment) and 6 months of follow-up
  The PSYRATS (Haddock et al, 1999; Gonzalez et al, 2003). This scale assess delusions in 6 items.

SECONDARY OUTCOMES:
Jumping to conclusions | baseline, 2 months (post-treatment) and 6 months of follow-up
  Three different computer tasks were used in the study. In Task 1, jars contained balls of two different colors; in one of them the proportion was 85 black versus 15 orange balls and in the other the ratio was reversed. Task 2 was the same as Task 1 but with a proportion of 60:40 in each jar. Finally, Task 3 was similar to Task 2 but instead of balls, the jars contained positive or negative comments with a proportion of 60:40. The patients had to decide which to jar belonged the extracted balls or comments. At all times the participants had information about the balls previously extracted, in order to control the effect of memory. The subjects could remove as many balls as needed to make their final decision (Garety et al., 2005). JTC was considered as taking a decision after extracting 1 or 2 balls.
BCIS. Beck Cognitive and Insight Scale | baseline, 2 months (post-treatment) and 6 months of follow-up. Moreover in the intervention group this scale was assessed at the end of each session
  The Beck Cognitive Insight Scale (BCSI; Beck et al., 2004; Gutierrez-Zotes et al., 2012) is a self-registering measure of 15 items which evaluates how the patients assess their own judgement. It has two dimensions; self-reflection (R) (9 items), and self-certainty (C) (6 items). A compound index of cognitive insight is obtained as the subtraction of self-certainty from self-reflection (R-C).
IPSAQ. Internal, Personal and Situational Attribution Questionnaire. | baseline, 2 months (post-treatment) and 6 months of follow-up.
  The scale assess the attributional style in 32 situations.
Hinking Task | baseline, 2 months (post-treatment) and 6 months of follow-up.
  The Scale assess Theory of Mind. For the porpouse of the study we selected 3 different situations in each assessment
TCI scale "Test de Creencias Irracionales" | baseline, 2 months (post-treatment) and 6 months of follow-up.
  This scale assess irrational beliefs in ten subscales:Need for acceptance by others, High self-expectations, blame, Intolerance to frustration, Worry and anxiety, Emotional irresponsibility, Avoidance of problems, dependency, helplessness, perfectionism.

OTHER OUTCOMES:
SFS "Social Functioning Scale" | baseline, 2 months (post-treatment) and 6 months of follow-up.
  This scale assess social functioning in people with psychotic disorders (Birchwood et al, 1990; Torres y Olivares, 2000).
Neuropsychological battery | baseline and 6 months of follow-up.
  A neuropsychological battery was included. The test included were WCST(Wisconsin Card Sorting Test, Bergs et al, 1948)measure of executive function; Test Stroop (Stroop, 1935) flexibility and inhibition of automatic responses; TMTA-B (Trail Making Test, Reitan, 1993) visual attention and task switching; CPT (Continous Performance Test, Conners 2000) this scale asses inattentiveness and impulsivity; TAVEC (Test Aprendizaje Verbal España Complutense, Benedet and Aleixandre 1998) this scale asses memory; WAIS (Weschler Adults Intelligence Scale, Wechsler 1955)subscales of digits and vocabulary.

CONTACTS AND LOCATIONS:
Overall Officials: Susana Ochoa, PhD, Principal Investigator — Parc Sanitari Sant Joan de Déu; Marisa Barrigón, PhD, Study Chair — Servicio Andaluz de Salud. Granada; Fermín González, Study Chair — Servicio Andaluz de Salud. Jaen; Isabel Ruiz, Study Chair — Servicio Andaluz de Salud. Málaga; Eva Grasa, Study Chair — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Esther Pousa, PhD, Study Chair — Corporacion Parc Tauli; Esther Lorente, PhD, Study Chair — Hospital Clínic de València; Ana Barajas, Study Chair — Centre d'Higiene Mental de les Corts; Jordi Cid, Study Chair — Institut d'Assistència Sanitària de Girona; Raquel López, MS, Study Chair — Parc Sanitari Sant Joan de Déu

REFERENCES:
- [Derived] Salas-Sender M, Lopez-Carrilero R, Barajas A, Lorente-Rovira E, Pousa E, Barrigon ML, Grasa E, Ruiz-Delgado I, Gonzalez-Higueras F, Cid J, Aznar A, Pelaez T, Birules I, Moritz S, The Spanish Metacognition Study Group, Ochoa S. Gender differences in response to metacognitive training in people with first-episode psychosis. J Consult Clin Psychol. 2020 Jun;88(6):516-525. doi: 10.1037/ccp0000468. Epub 2019 Dec 19. PMID 31855037